CLINICAL TRIAL: NCT04020484
Title: A Live-Online Mindfulness-based Intervention for Families of Children With Epilepsy: Making Mindfulness Matter© Randomized Control Trial
Brief Title: Making Mindfulness Matter© in Children With Epilepsy
Acronym: M3Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6558
Record Dates: First submitted 2019-05-24; First posted 2019-07-16 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy in Children; Mindfulness; Quality of Life

STUDY DESIGN:
Intervention Model Description: This is a parallel, partially nested randomized controlled trial (RCT) comparing two arms: intervention (M3) and treatment-as-usual (i.e. wait-list control). Participants will be randomized 1:1 into the intervention or control arm. This study will not interfere with patients' clinical care. The intervention will be delivered online to groups of 4-8 on a rolling basis to minimize wait-times and allow for timely access to the intervention for the waitlist controls. We believe this strategy is very important to increase the odds that families will decide to participate in the study. Sample size calculations showed that 76 child-parent dyads will be required (38 intervention, 38 control), and to account for a liberal 24% attrition rate, 100 child-parent dyads will be recruited.
Who Masked: Participant, Care Provider
Masking Description: Blinding of participants and program facilitators (i.e. the staff delivering the M3 program) will be difficult to completely achieve given the nature of the intervention. The investigators will attempt to ameliorate bias by explaining to participants and program facilitators that the study is interested in evaluating the intervention to be given to all participants, however, in planning the logistics of the intervention, some participants will receive the intervention in the very near future, whereas others will receive the intervention in approximately 12 weeks. In so doing, the investigators hope to eliminate any biases associated with the participants' and program facilitators' perception or biases of being assigned to the treatment or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Child-parent dyads will undergo a standardized 8-week course of Making Mindfulness Matter© (M3). The program will be delivered online using live, interactive sessions to groups of 4 to 8, for 1.5 hours each week for the parent group and 1 hour each week for the child group. Children and parents will attend separate on-line sessions and at the end of each child session, the parent will be asked to join their child on-line for a shared mindful exercise. Once 4 to 8 dyads are assigned to the intervention group, participants will be given the baseline questionnaires and start the intervention in the following week.
  Interventions: Behavioral: Making Mindfulness Matter© (M3)
- Waitlist Control (Other): Child-parent dyads randomized to the control arm will continue treatment as usual. Once 4 to 8 dyads are assigned to the control group, participants will be given the baseline questionnaires, They will complete the Baseline and Immediate Follow-up questionnaire at comparable times to families in the intervention arm; they will not complete the Extended Follow-up questionnaire. These dyads will be provided with the intervention at the next scheduled session; the goal is to provide the intervention to controls as soon as possible to avoid differential attrition between the intervention and control arm. During the intervention sessions, they will complete all feasibility surveys pertaining to the intervention and their satisfaction with each intervention session.
  Interventions: Behavioral: Making Mindfulness Matter© (M3)

INTERVENTIONS:
Behavioral: Making Mindfulness Matter© (M3) — Making Mindfulness Matter© (M3) is an interactive online parent and child program that incorporates mindful awareness, social-emotional learning skills, neuroscience, and positive psychology. This program was modelled after the school-based MindUP™ program for use in the community and augmented to integrate a parent component. M3E is a facilitator-led program that integrates attitudes, skills, and behaviours related to mindfulness and social-emotional learning (SEL). During the 8-week concurrent parent and child manualized program, parents learn the same core principles as children: how our brains work, stress and the brain, mindful breathing, mindful sensing, mindful movement, perspective taking, optimism, and gratitude/acts of kindness.
  Other Names: M3E

SUMMARY:
Epilepsy is a debilitating condition characterized by spontaneous, unprovoked seizures. Up to 80% of children with epilepsy (CWE) may face cognitive, psychiatric, and/or behavioral comorbidities with significant unmet mental health needs. Mindfulness-based interventions may provide an ideal vector to target unmet mental healthcare needs in patients with epilepsy and their families. The investigators propose the Making Mindfulness Matter© (M3) program as an intervention to improve health related quality of life and mental-health for CWE and their parents. M3 is live-online parent and child program that incorporates mindful awareness, social-emotional learning skills, neuroscience, and positive psychology. This pilot RCT is needed to refine the implementation of the intervention to families with a child with epilepsy, and collect information pertaining to the feasibility and effectiveness of the intervention in preparation for a subsequent multi-centred trial across Canada. Note: Due to COVID-19, the format has been modified for online delivery (from community-based) and the intervention has been restarted.

DETAILED DESCRIPTION:
Recognizing that medical management for chronic illness such as epilepsy does not address the stress and co-occurring psychological issues experienced by many patients, mindfulness-based interventions have been increasingly utilized. Mindfulness-based interventions are effective, well-validated interventions for several adult outcomes including physical and mental health, social and emotional well-being, and cognition. Meta-analyses report overall medium effect sizes of 0.50 to 0.59 across these outcomes. In a recent Cochrane review of psychological interventions for people with epilepsy, three studies specifically examined mindfulness-based techniques for adults with epilepsy and determined positive outcomes on mental health, HRQOL and seizure outcomes. There has been far less research on mindfulness with children and youth than in adults; studies that have been done have been plagued with methodological limitations including small numbers, lack of randomization or control groups. However, evidence to-date indicates that mindfulness interventions for children and youth are feasible, accepted and enjoyed by participants. The few well conducted studies on mindfulness interventions in children without physical health issues have reported reduced symptoms of anxiety, depression, and stress, reduced maladaptive coping and rumination, and improved behavioural and emotional self-regulation and focus. Furthermore, a recent systematic review and meta-analysis found that mindfulness interventions were three times more effective in alleviating psychological symptoms among children with clinically diagnosed psychological disorders (such as anxiety, learning disability and externalizing disorders), compared with healthy controls. This suggests that mindfulness interventions may be particularly relevant for those with clinical levels of psychological disorders, a particularly relevant finding for our study given that children with epilepsy experience greater levels of depression, anxiety, learning disability and behavioural comorbidities.

In addition to the benefits of programs that deliver mindfulness interventions directly to children, programs that target parents and parents appear to be effective in improving parental functioning and in turn, promote child outcomes. Furthermore, studies are indicating that mindfulness-based interventions for parents of children with chronic issues (attention deficit hyperactivity disorder, developmental delays, autism) are effective for lessening parental stress and mental health problems. Improvements in parent-child relationship and improved youth behaviour management have also been found.

Neither the Cochrane review on the impact of psychological treatments for people with epilepsy, nor a recent systematic review on mindfulness interventions in youth found studies investigating mindfulness management techniques for CWE. Despite the paucity of studies of mindfulness interventions in childhood epilepsy, there is converging evidence to suggest studying a mindfulness-based intervention in children and families with epilepsy is warranted. There is research pointing to the effectiveness of mindfulness-based interventions on psychological symptoms in adults and children, especially in those with relevant clinical issues similar to CWE. The investigators believe the M3 program is ideally suited for use with CWE and their parents for a number of reasons. The program was developed from the validated, widely used, and successful Mind UP program for use in the community and augmented to integrate a parent component, and has been shown to be successful in our cohort of young children and their parents facing adversity. Importantly, M3 is suitable for children as young as 4 years of age, which is particularly important as evidence to date suggests that early identification and treatment of epilepsy comorbidities is essential as there may be a window of opportunity for early intervention in some children. Interventions must be implemented early before problems become entrenched and interfere with the development of basic cognitive, behavioral, and social skills crucial for long-term educational, vocational, and interpersonal adaptation. The low-cost, interactive online group delivery and facilitation by non-clinician staff also allows the program to be scalable to communities across Canada and increases its likely sustainability.

ELIGIBILITY:
No age restriction on parent participating in parent/child dyad

Inclusion Criteria:

1. Children aged 4 to 10 years diagnosed with epilepsy a minimum of 6 months ago, as per the International League Against Epilepsy (ILAE) 2014 operational definition*
2. Children have reasonable comprehension of spoken language and can follow simple instructions
3. Children with epilepsy and their parents** are willing to attend all intervention sessions
4. Children with epilepsy and parents have an adequate understanding of English

   * Operational (practical) clinical definition of epilepsy (Fisher et al. 2014):

     1. At least two unprovoked (or reflex) seizures occurring>24 h apart, or
     2. One unprovoked (or reflex) seizure and a probability of further seizures similar to the general recurrence risk (at least 60%) after two unprovoked seizures, occurring over the next 10 years, or
     3. Diagnosis of an epilepsy syndrome

        * Parents: refers to parent or guardian self-identifying as most responsible for child's day-to-day care

Exclusion criteria are:

1. Progressive or degenerative neurological disorder;
2. Other major co-morbid non-neurological disorders (e.g. cystic fibrosis, Crohn's disease, diabetes, renal failure);
3. Concurrent enrollment in other intervention trials
4. Child or parent regularly practice complementary health interventions such as meditation
5. Scheduled to undergo epilepsy surgery during study period

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of Making Mindfulness Matter© (M3) as a family treatment for children with epilepsy and their parents | Throughout the study enrollment period and over the 8 weeks of intervention.
  The investigators will track the number of patients contacted, response rate, attrition and reasons for non-participation and attrition. At the start of each session, parents will complete a one-page (12-item) semi-structured questionnaire evaluating treatment fidelity, at home utilization of M3 skills. At the end of each session, parents will complete an overall feedback form on the intervention. Facilitators will complete a two-page questionnaire providing feedback on the session. At the start and end of the M3 program, children will be asked to complete a feeling face questionnaire rated on a 3-point scale about topics discussed in the group such as how our brain works when upset and what is mindfulness.

SECONDARY OUTCOMES:
Effect of M3 on Health Related Quality of Life of children with epilepsy | baseline, 8 weeks, 17 weeks
  The Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55) is a 55-item measure that emphasizes a functional approach to quality of life. QOLCE-55 generates an overall quality of life score, and four subscale scores: cognitive, emotional, social and physical functioning. Scores range from 0 to 100, with higher scores indicative of better quality of life.
  Although the QOLCE is a widely used HRQOL scale, no study has calculated the minimum clinically important difference (MCID). To calculate the MCID for the QOLCE, the Patient Centred Global Ratings of Change will be used, a 5-item scale where respondents indicate the amount of change relative to baseline. Rating from -7 (much worse) through 0 (no change) to +7 (much better). This information will allow us to calculate the MCID for the QOLCE-55, and thereby identify the proportion of patients who experience a clinically meaningful change following intervention.
Effect of M3 on Health Related Quality of Life of parents | baseline, 8 weeks, 17 weeks
  The Short Form Health Survey (SF12v2), a 12-item self-reported measure evaluating physical and mental health components of health-related quality of life over the past 4 weeks will be used. The measures generates two composite scales relating to the physical and mental health components of health related quality of life. This measure is the most frequently used patient reported outcome in clinical trials, and has been used most frequently in studies evaluating quality of life of parents of children with epilepsy.
Does M3 have a positive effect on children's externalizing problems | baseline, 8 weeks, 17 weeks
  Behavior Assessment System for Children (BASC-3) 139-175-item comprehensive scale evaluating children's adaptive and problem behaviors in community and home settings. The BASC composite scale 'externalizing problems' will be used. Persons with T-score above 59 in a given scale are categorized as 'at-risk' for that domain.
Does M3 have a positive effect on children's internalizing problems | baseline, 8 weeks, 17 weeks
  Behavior Assessment System for Children (BASC-3) 139-175-item comprehensive scale evaluating children's adaptive and problem behaviors in community and home settings. The BASC composite scale 'internalizing problems' will be used. Persons with T-score above 59 in a given scale are categorized as 'at-risk' for that domain.
Does M3 have a positive effect on children's adaptive skills | baseline, 8 weeks, 17 weeks
  Behavior Assessment System for Children (BASC-3) 139-175-item comprehensive scale evaluating children's adaptive and problem behaviors in community and home settings. The BASC composite scale 'adaptive skills' will be used. Persons with T-score above 59 in a given scale are categorized as 'at-risk' for that domain.
Does M3 have a positive effect on children's executive function | baseline, 8 weeks, 17 weeks
  Behavioral Rating Inventory of Executive Function 2 (BRIEF) 86-item scale measuring parent-rated executive function and self-regulation in children. Generates a global executive composite, cognitive regulation index, emotion regulation index, behavior regulation index. Persons with T-score above 60 in a given scale are categorized as 'at-risk' for that domain.
Does M3 have a positive effect on children's severity of epilepsy | baseline, 8 weeks, 17 weeks
  Parents will rate the child's epilepsy severity using the Global assessment of the severity of epilepsy (GASE), a single item measure scale measured on a 7-point Likert type scale. Seizure frequency will be rated by parents through two questions asking the number of seizures and number of seizure-free days in the past 30 days.
Does M3 have a positive effect on parents' depression | baseline, 8 weeks, 17 weeks
  Center for Epidemiological Studies Depression Scale (CES-D) 20-item scale evaluating the level of depressive symptoms, and is one of the most widely used instruments in the field of psychiatric epidemiology. Generates an overall score for depressive symptoms, with scores above 16 indicative of risk for depression.
Does M3 have a positive effect on parents' anxiety | baseline, 8 weeks, 17 weeks
  Generalized Anxiety Disorder 7-item (GAD-7) scale evaluating generalized anxiety. Generates an overall anxiety score, with scores above 10 indicative of moderate-severe anxiety.
Does M3 have a positive effect on parents' stress | baseline, 8 weeks, 17 weeks
  Parenting Stress Index 4 - short form 36-item scale that helps identify sources of stress. Focused on three major domains of stress: child characteristics, parent characteristics, and situational/demographic factors. A summary and 3 subscale (Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child) scores are generated. Scores in the 81st percentile or higher are indicative of high stress.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Nixon Speechley, Ph.D, Principal Investigator — Western University; Klajdi Puka, Ph.D, Principal Investigator — CAMH; Karen Bax, Ph.D, Principal Investigator — Western University
Locations (1):
- Epilepsy Southwestern Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puka K, Bax K, Andrade A, Devries-Rizzo M, Gangam H, Levin S, Nouri MN, Prasad AN, Secco M, Zou G, Speechley KN. A live-online mindfulness-based intervention for children living with epilepsy and their families: protocol for a randomized controlled trial of Making Mindfulness Matter(c). Trials. 2020 Nov 11;21(1):922. doi: 10.1186/s13063-020-04792-3. PMID 33176853